CLINICAL TRIAL: NCT03187080
Title: Evaluating the Use of Enhanced Recovery Strategies and Paravertebral Block in Elective Breast Reduction and Breast Augmentation
Brief Title: Enhanced Recovery Strategies in Elective Breast Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: per Research Hold
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-1388; A539730 (Other: UW Madison); SMPH\SURGERY\DENT&P SRG (Other: UW Madison); Protocol Version 4/9/2021 (Other: UW Madison)
Record Dates: First submitted 2017-06-01; First posted 2017-06-14 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pain, Acute; Nausea; Vomiting, Postoperative; Opioid Use; Satisfaction
MeSH Terms: conditions — Acute Pain; Nausea; Postoperative Nausea and Vomiting; Personal Satisfaction | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: There are four serial aims of this study. The overarching goal is to prospectively assess the use of PVB as an adjunct for postoperative pain control both alone and in the setting of related ERABS strategies in elective breast surgery (both breast reduction and breast augmentation, two of the most common non-oncologic breast operations performed in an ambulatory setting). The methodologies used to assess postoperative pain, the set of collective ERABS strategies, the potential risks and benefits of study participation, and the inclusion/exclusion criteria will be the same in the groups studying breast reduction and those studying breast augmentation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be blinded as to which treatment arm within their group that they are allocated. The surgery team including the surgeon (PI) and resident will be blinded as well. Anesthesiologists will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1 Arm A (Experimental): Breast reduction with Paravertebral block using local anesthetic.
  Interventions: Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline; Drug: Paravertebral block using local anesthetic
- Group 1 Arm B (Sham Comparator): Breast reduction with Sham paravertebral block using saline.
  Interventions: Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline; Procedure: Sham paravertebral block using saline
- Group 2 Arm A (Experimental): Breast augmentation with Paravertebral block using local anesthetic.
  Interventions: Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline; Drug: Paravertebral block using local anesthetic
- Group 2 Arm B (Sham Comparator): Breast augmentation with Sham paravertebral block using saline.
  Interventions: Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline; Procedure: Sham paravertebral block using saline
- Group 3 Arm A (Experimental): Breast reduction with Enhanced recovery after breast surgery (ERABS) strategies.
  Interventions: Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline; Other: Enhanced recovery after breast surgery (ERABS) strategies
- Group 3 Arm B (No Intervention): Breast reduction, standard perioperative management.
- Group 4 Arm A (Experimental): Breast augmentation with Enhanced recovery after breast surgery (ERABS) strategies.
  Interventions: Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline; Other: Enhanced recovery after breast surgery (ERABS) strategies; Drug: Paravertebral block using local anesthetic
- Group 4 Arm B (No Intervention): Breast augmentation, standard perioperative management.

INTERVENTIONS:
Procedure: Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline — Paravertebral block (PVB) will be performed in the standard fashion using an out-of-plane ultrasound approach by an anesthesiologist with appropriate training in regional anesthesia. Landmarks on the patient will be identified. The skin will be sterilized. The intended target (paravertebral space) will be located using an ultrasound. A Pajunk UniPlex NanoLine needle will be inserted. A syringe filled with sterile saline (used for hydrodissection) connected to a syringe of 0.25% bupivacaine with 2.5 mcg/mL of epinephrine will be connected to the Pajunk needle and used for injection. The needle will be advanced toward and through the superior costotransverse ligament or internal intercostal membrane. Once through the ligament, the pleura will be seen deflecting anteriorly with the hydrodissection. Negative aspiration will be confirmed, and the local anesthetic will be injected into the paravertebral space.
  Arms: Group 1 Arm A; Group 1 Arm B; Group 2 Arm A; Group 2 Arm B; Group 3 Arm A; Group 4 Arm A
Other: Enhanced recovery after breast surgery (ERABS) strategies — For comparing ERABS strategies to current standard of care, the following perioperative strategies will be utilized:
  * Standardized written information given preoperatively.
  * Allow clear liquids for up to 2 hours prior to arrival at the surgery center.
  * Use paravertebral block to augment postoperative pain control.
  * Standardized multimodal analgesic regimen
  * Antiemetics
  * Easily accessible call-in or walk-in postop care/support
  The proposed strategies differ from standard of care in the following ways:
  * PVB is less commonly used in elective surgery.
  * Patients do not eat or drink after midnight.
  * There is no standardized preoperative information packet.
  * Anesthetic/intraoperative analgesic and antiemetic regimen varies between providers.
  Arms: Group 3 Arm A; Group 4 Arm A
Procedure: Sham paravertebral block using saline — Paravertebral block (PVB) will be performed in the standard fashion using an out-of-plane ultrasound approach by an anesthesiologist with appropriate training in regional anesthesia. Landmarks on the patient will be identified. The skin will be sterilized. The intended target (paravertebral space) will be located using an ultrasound. A Pajunk UniPlex NanoLine needle will be inserted. A syringe filled with sterile saline (used for hydrodissection) connected to a syringe of sterile saline will be connected to the Pajunk needle and used for injection. The needle will be advanced toward and through the superior costotransverse ligament or internal intercostal membrane. Once through the ligament, the pleura will be seen deflecting anteriorly with the hydrodissection. Negative aspiration will be confirmed, and the local anesthetic will be injected into the paravertebral space.
  Arms: Group 1 Arm B; Group 2 Arm B
Drug: Paravertebral block using local anesthetic — Use of local anesthetic (0.25% bupivacaine) that is *NOT* an experimental drug but will be used as part of the paravertebral block to provide local anesthetic. This will not be given to those in the sham block groups.
  Arms: Group 1 Arm A; Group 2 Arm A; Group 4 Arm A

SUMMARY:
Postoperative pain, nausea, and vomiting are frustrating sequelae of elective breast surgery. Poorly managed postoperative pain can lead to increased opioid use, increased postoperative nausea and vomiting (PONV), delayed return to work and usual activities, unplanned hospital admissions, surgical complications, and patient dissatisfaction. In light of the growing opioid epidemic in the United States, any intervention that potentially minimizes opioid use may have meaningful individual and societal impact. In patients undergoing breast reduction and breast augmentation surgery, multiple techniques for managing postoperative pain are used commonly. One such technique is the use of a paravertebral block (PVB), which is a method of injecting local anesthesia into the area surrounding the spinal nerves in order to decrease sensation and pain in the chests and breasts in the setting of breast surgery. PVB is generally used concomitantly with standard multimodal perioperative pain management including cool compress, non-steroidal anti-inflammatories (NSAIDs), acetaminophen, and opioids. All of these pain management strategies are used at the University of Wisconsin and are considered standard of care for breast surgery nationwide.

The overall purpose of this study is to evaluate interventions that aim to optimize pain control, minimize the risk of PONV, and improve recovery after elective breast surgery. The investigators will do this by (1) Comparing PVB with standard pain management strategies in patients undergoing planned breast reduction and breast augmentation, and (2) Comparing "enhanced recovery after surgery" (ERAS) strategies to standard of care for patients undergoing planned breast reduction and breast augmentation. This will be studied using pain assessments, validated surveys, medication logs, and review of medical records.

DETAILED DESCRIPTION:
Bilateral breast reduction and bilateral breast augmentation are both routine plastic surgery procedures commonly performed on an outpatient basis. While patient satisfaction following these procedures is high, postoperative pain management can be challenging, resulting in decreased patient satisfaction, delayed recovery including delayed return to work and daily activities, increased opioid pain medication requirements and occasionally unplanned hospital admissions, surgical complications, and increased cost of care.

PVB is a common procedure used for analgesia in breast surgery in combination with multimodal perioperative pain regimens, though its use has not been formally studied in a prospective fashion. To date, no prospective, randomized, blinded study has been performed to evaluate the efficacy of PVB on perioperative pain management in this patient population.

The overarching goal of this study is to evaluate the safety and efficacy of PVB alone, as well as in conjunction with a global set of perioperative enhanced recovery strategies in elective breast surgery. The investigators hypothesize that the use of such strategies will improve the patient experience of breast reduction and augmentation beyond the current standard of care.

There are four serial aims of this study. The overarching goal of the study is to prospectively assess the use of PVB as an adjunct for postoperative pain control both alone and in the setting of related ERABS strategies in elective breast surgery (both breast reduction and breast augmentation, two of the most common non-oncologic breast operations performed in an ambulatory setting). The methodologies used to assess postoperative pain, the set of collective ERABS strategies, the potential risks and benefits of study participation, and the inclusion/exclusion criteria will be the same in the groups studying breast reduction and those studying breast augmentation.

Following completion of all 4 groups, the investigators will be able to assess the impact of PVB alone as well as the impact of ERABS strategies in both breast reduction and breast augmentation.

The primary aim in all four groups in this study is to evaluate postoperative pain scores in patients receiving either paravertebral block or ERABS strategies compared to patients who do not receive these interventions. Additional outcomes include use of analgesic and antiemetic medication, development of PONV, time to discharge, patients' assessment of quality of recovery as determined by a validated survey and overall patient satisfaction.

Group 1: To prospectively determine the effect of PVB on perioperative pain and postoperative recovery following breast reduction. Patient-reported pain assessments (including a numeric rating scale) will be used to evaluate the primary endpoint (pain scores on postoperative day 1 (POD1)) as well as additional outcome measures of pain scores in recovery and at 1 week post-surgery. To determine the effect of PVB on secondary endpoints of this study, analgesic and antiemetic medication use will be calculated, average time (minutes) spent in the Post Anesthesia Care Unit (PACU), average time (minutes) spent in Phase 2, and total time (minutes) between the end of the operation and discharge to home will be compared, the occurrence of unplanned hospital admission will be evaluated, PONV assessed, overall satisfaction, patients' assessment of quality of recovery as determined by a validated survey, and complications documented. This data will be obtained through review of medical records, surveys, and postoperative diaries.

Patients electing to undergo breast reduction will be invited to participate in the study at their preoperative visit. All patients choosing to take part in the study will be consented prior to their procedure. The study participants will be randomized to one of two arms within each Group using block randomization. Details of the allocated group will be written on a piece of paper and placed inside sealed, opaque, and sequentially numbered, envelopes. Block randomization will be performed using a computer-generated number list and an Excel spreadsheet template. Block randomization will ensure equal numbers of subjects in each group. Either the anesthesiologist or the surgical team will open the envelope when the patient presents to UW Transformations Surgery Center or Madison Surgery Center (MSC) the day of surgery. The subject will be randomized to receive either (a) standard postoperative nausea and pain control as well as a sham superficial injection of normal saline or (b) PVB in addition to standard postoperative nausea and pain control. PVB and sham superficial injections of normal saline will be performed by a trained anesthesiology provider and will be performed in the routine manner. Surgery will take place in the usual fashion and participants will receive standard of care for pain and nausea control.

Following surgery, patients will be assessed for postoperative pain, nausea and vomiting. Assessment for postoperative pain will consist of a validated pain score survey administered prior to transfer to phase II postoperatively, on POD1, and at their one-week postoperative visit. Participants will also be asked to record, using a postoperative diary/log, when they take postoperative analgesics and antiemetics, which medications are taken, and quantity of medication taken. This will also be reviewed both in the medical record and upon discussion with the participant at the postoperative visits. Assessment of the time spent in the recovery room, time spent in Phase 2 of recovery, and time to discharge from the hospital (total time between the end of surgery to discharge from hospital), will be obtained via review of the medical record. At the first postoperative visit, participants will undergo a routine interview that includes discussion of their pain control, analgesic and antiemetic use, recovery process, and overall satisfaction. The medical record will be reviewed for any unplanned postoperative hospital readmissions related to the surgery.

Group 2: To prospectively determine the effect of PVB on perioperative pain and postoperative recovery following breast augmentation. Patient-reported pain assessments (including a numeric rating scale) will be used to evaluate the primary endpoint (pain scores on postoperative day 1 (POD1)) as well as additional outcome measures of pain scores in recovery and at 1 week post-surgery. To determine the effect of PVB on secondary endpoints of this study, analgesic and antiemetic medication use will be calculated, average time (minutes) spent in the PACU, average time (minutes) spent in Phase 2, and total time (minutes) between the end of the operation and discharge to home will be compared, the occurrence of unplanned hospital admission will be evaluated, PONV assessed, overall satisfaction, patients' assessment of quality of recovery as determined by a validated survey, and complications will be documented. This data will be obtained through review of medical records, surveys, and postoperative diaries.

The procedures will be the same as those described for Group 1, except patients will be undergoing planned breast augmentation.

Groups 3 and 4: To prospectively compare the standard of care for ambulatory breast surgery to "fast track" (also known as "enhanced recovery") strategies for breast surgery by assessing pain scores, pain medication and antiemetic use, development of nausea/vomiting, time to discharge, and patient satisfaction.

For the third serial Group in the study, patients electing to undergo breast reduction surgery will be invited to participate in the study at their preoperative visit. For the fourth Group in the study, all procedures will be the same as described in this section, but the patients will be undergoing breast augmentation surgery (not breast reduction). All patients choosing to take part in the study will be consented prior to their procedure. The study participants will be randomized, using block randomization, a computer-generated randomization template, and sealed, numbered, and opaque envelopes, to either receive (a) perioperative pain, nausea, and recovery strategies as part of our Enhanced Recovery after Breast Surgery (ERABS) protocol, or (b) perioperative instructions, anesthesia and medications as per our institution's current standard of care for elective breast reduction or breast augmentation.

Validated pain assessments will be used to evaluate the primary endpoint (pain scores on postoperative day 1 (POD1)) as well as additional outcome measures of pain scores in recovery and at 1 week post-surgery. To determine the effect of PVB on secondary endpoints of this study, analgesic and antiemetic medication use will be calculated, average time (minutes) spent in the PACU, average time (minutes) spent in Phase 2, and total time (minutes) between the end of the operation and discharge to home will be compared, and the occurrence of unplanned hospital admission will be evaluated, occurrence of PONV assessed, assessment of recovery, overall satisfaction, and complications documented. This data will be obtained through review of medical records, questionnaires, and postoperative diaries.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to and greater than 18 years.
* Medically cleared to undergo elective breast surgery (including associated anesthesia) at UW Transformations Surgery Center or Madison Surgery Center (MSC).
* Undergoing bilateral breast augmentation or bilateral breast reduction by the PI (Dr. Venkat Rao).

Exclusion Criteria:

* Minors or under the age of 18
* Pregnant or breast feeding women
* Incarcerated women
* Males
* Individuals unable to give consent due to another condition such as impaired decision-making capacity.
* Women who take opioid pain medications on a regular basis prior to surgery.
* Women with a history of opioid abuse and/or dependence.
* Women who, based on anesthesiologist discretion, are not candidates for paravertebral block.
* Women with BMI >35
* Women with a diagnosis of obstructive sleep apnea who are noncompliant with their treatment (e.g. CPAP use).
* Women with a history of bleeding disorders precluding safe paravertebral block.
* Women on anticoagulation therapy who have not held their anticoagulation as recommended by their surgeon or anesthesiologist.
* Women with a history of infection at the site of paravertebral block.
* Women not medically cleared for surgery at Transformations or MSC and thus would not be undergoing surgery at Transformations or MSC. This would include women with sepsis/bacteremia, significant valvular disorders or heart conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkat K Rao, MD, MBA, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonde C, Khorasani H, Eriksen K, Wolthers M, Kehlet H, Elberg J. Introducing the fast track surgery principles can reduce length of stay after autologous breast reconstruction using free flaps: A case control study. J Plast Surg Hand Surg. 2015;49(6):367-71. doi: 10.3109/2000656X.2015.1062387. Epub 2015 Jul 10. PMID 26161838
- [Background] Davis GM, Ringler SL, Short K, Sherrick D, Bengtson BP. Reduction mammaplasty: long-term efficacy, morbidity, and patient satisfaction. Plast Reconstr Surg. 1995 Oct;96(5):1106-10. PMID 7568486
- [Background] Parikh RP, Sharma K, Guffey R, Myckatyn TM. Preoperative Paravertebral Block Improves Postoperative Pain Control and Reduces Hospital Length of Stay in Patients Undergoing Autologous Breast Reconstruction after Mastectomy for Breast Cancer. Ann Surg Oncol. 2016 Dec;23(13):4262-4269. doi: 10.1245/s10434-016-5471-1. Epub 2016 Aug 3. PMID 27489056
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Anderson AD, McNaught CE, MacFie J, Tring I, Barker P, Mitchell CJ. Randomized clinical trial of multimodal optimization and standard perioperative surgical care. Br J Surg. 2003 Dec;90(12):1497-504. doi: 10.1002/bjs.4371. PMID 14648727
- [Background] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Arsalani-Zadeh R, ElFadl D, Yassin N, MacFie J. Evidence-based review of enhancing postoperative recovery after breast surgery. Br J Surg. 2011 Feb;98(2):181-96. doi: 10.1002/bjs.7331. PMID 21104705
- [Background] Kairaluoma PM, Bachmann MS, Korpinen AK, Rosenberg PH, Pere PJ. Single-injection paravertebral block before general anesthesia enhances analgesia after breast cancer surgery with and without associated lymph node biopsy. Anesth Analg. 2004 Dec;99(6):1837-1843. doi: 10.1213/01.ANE.0000136775.15566.87. PMID 15562083
- [Background] Dabbagh A, Elyasi H. The role of paravertebral block in decreasing postoperative pain in elective breast surgeries. Med Sci Monit. 2007 Oct;13(10):CR464-7. PMID 17901854
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from October 2017 to June 2021. Research was put on Divisional Hold in January 2022. May 2024 determination was made to close the study.
Groups:
- Group 1 Arm A: Breast reduction with Paravertebral block using local anesthetic.
  Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline: Paravertebral block (PVB) will be performed in the standard fashion using an out-of-plane ultrasound approach by an anesthesiologist with appropriate training in regional anesthesia.
  Paravertebral block using local anesthetic: Use of local anesthetic (0.25% bupivacaine) that is *NOT* an experimental drug but will be used as part of the paravertebral block to provide local anesthetic. This will not be given to those in the sham block groups.
- Group 1 Arm B: Breast reduction with Sham paravertebral block using saline.
  Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline: Paravertebral block (PVB) will be performed in the standard fashion using an out-of-plane ultrasound approach by an anesthesiologist with appropriate training in regional anesthesia.
- Group 2 Arm A: Breast augmentation with Paravertebral block using local anesthetic.
  Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline: Paravertebral block (PVB) will be performed in the standard fashion using an out-of-plane ultrasound approach by an anesthesiologist with appropriate training in regional anesthesia.
  Paravertebral block using local anesthetic: Use of local anesthetic (0.25% bupivacaine) that is *NOT* an experimental drug but will be used as part of the paravertebral block to provide local anesthetic. This will not be given to those in the sham block groups.
- Group 2 Arm B: Breast augmentation with Sham paravertebral block using saline.
  Paravertebral block procedure using either local anesthetic (0.25% bupivacaine) or sterile saline: Paravertebral block (PVB) will be performed in the standard fashion using an out-of-plane ultrasound approach by an anesthesiologist with appropriate training in regional anesthesia.
- Group 3 Arm A: Breast reduction with Enhanced recovery after breast surgery (ERABS) strategies.
  Enhanced recovery after breast surgery (ERABS) strategies: For comparing ERABS strategies to our current standard of care, we will utilize the following perioperative strategies:
  * Standardized written information given preoperatively.
  * Allow clear liquids for up to 2 hours prior to arrival at the surgery center.
  * Use paravertebral block to augment postoperative pain control.
  * Standardized multimodal analgesic regimen
  * Antiemetics
  * Easily accessible call-in or walk-in postop care/support
  The proposed strategies differ from standard of care in the following ways:
  * PVB is less commonly used in elective surgery.
  * Patients do not eat or drink after midnight.
  * There is no standardized preoperative information packet.
  * Anesthetic/intraoperative analgesic and antiemetic regimen varies between providers.
- Group 4 Arm A: Breast augmentation with Enhanced recovery after breast surgery (ERABS) strategies.
  Enhanced recovery after breast surgery (ERABS) strategies: For comparing ERABS strategies to our current standard of care, we will utilize the following perioperative strategies:
  * Standardized written information given preoperatively.
  * Allow clear liquids for up to 2 hours prior to arrival at the surgery center.
  * Use paravertebral block to augment postoperative pain control.
  * Standardized multimodal analgesic regimen
  * Antiemetics
  * Easily accessible call-in or walk-in postop care/support
  The proposed strategies differ from standard of care in the following ways:
  * PVB is less commonly used in elective surgery.
  * Patients do not eat or drink after midnight.
  * There is no standardized preoperative information packet.
  * Anesthetic/intraoperative analgesic and antiemetic regimen varies between providers.
Period: Overall Study
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Started | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
Completed | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study Terminated Early
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B | Total
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (21.7) |  |  |  | 31.0 (17.5) |  | 26.6 (20.1) |  | 34.9 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 |  |  |  | 16 |  | 32 |  | 113
  Male | 0 |  |  |  | 0 |  | 0 |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 65 |  |  |  | 16 |  | 32 |  | 113
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — weight in kilograms divided by the square of height in meters (kg/m^2)
  kg/m^2 | 32.6 (4.7) |  |  |  | 32.8 (5.4) |  | 24.4 (2.8) |  | 30.3 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Pain Scores, Rated by Patient on 0-10 Scale
Description: Our primary outcome of interest is self-reported pain (0-10 visual analog scale) on post-operative day 1 (POD1). Higher scores indicates higher levels of pain.
Time Frame: Postoperative day 1
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
score on a scale | 5.8 (2.3) |  |  |  | 5.9 (1.9) |  | 6.7 (1.8) |

2. Secondary Outcome: Numerical Pain Scores, Rated by Patient on 0-10 Scale
Description: Pain scores in Post Anesthesia Care Unit (PACU) / recovery area. Pain scored from 0-10 where higher scores indicates higher levels of pain.
Time Frame: Day of surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
score on a scale | 4.7 (2.5) |  |  |  | 5.4 (3.3) |  | 4.5 (2.3) |

3. Secondary Outcome: Time Spent in Each Phase of Care Prior to Discharge
Description: Time spent in recovery after surgery in the PACU and Phase II (the area of recovery that patients transition to between PACU and discharge)
Time Frame: Day of surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
minutes
  PACU | 42 (38) |  |  |  | 25 (17) |  | 28 (15) |
  Phase II | 92 (58) |  |  |  | 64 (43) |  | 99 (55) |

4. Secondary Outcome: Time to Discharge to Home
Description: Time between conclusion of surgery and discharge from the surgery center
Time Frame: Day of surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
minutes | 127 (78) |  |  |  | 127 (67) |  | 89 (56) |

5. Secondary Outcome: Analgesic Requirements Reported as the Number of Participants Who Were Still Taking Medications Post-Operatively Day 7
Time Frame: 1 week after surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
Participants
  Oxycodone | 0 |  |  |  | 1 |  | 1 |
  Tylenol | 2 |  |  |  | 2 |  | 4 |
  Ibuprofen | 2 |  |  |  | 2 |  | 3 |

6. Secondary Outcome: Post-operative Nausea and Vomiting (Subjective Report) Measured as the Mean Incidence Reported Post-Operatively Day 7
Description: Occurrence of nausea and vomiting after surgery
Time Frame: 1 week after surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
events per week | 3.2 (1.6) |  |  |  | 0.45 (1.0) |  | 1.0 (1.1) |

7. Secondary Outcome: Anti-emetic Requirements Measured as Number of Participants Taking Anti-nausea Medication Post-Operatively Day 7
Description: Use of anti-nausea mediation postoperatively
Time Frame: 1 week after surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
Participants | 0 |  |  |  | 0 |  | 0 |

8. Secondary Outcome: Patients' Assessment of Perceived Quality of Recovery Using Modified Quality of Recovery Survey (MQOR-40)
Description: Patients' assessment of quality of recovery using validated 'quality of recovery 40' survey. This survey is scored from 1-5 where higher scores indicate better quality of recovery.
Time Frame: 1 week after surgery
Population: Study was terminated early, participants not enrolled in all planned arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
Number analyzed (Participants) | 65 | 0 | 0 | 0 | 16 | 0 | 32 | 0
score on a scale | 3.3 (1.6) |  |  |  | 2.3 (2.1) |  | 2.3 (2.0) |

ADVERSE EVENTS:
Time Frame: up to 1 week post op
Description: study terminated early, participants not enrolled into all arms
Arm/Group | Group 1 Arm A | Group 1 Arm B | Group 2 Arm A | Group 2 Arm B | Group 3 Arm A | Group 3 Arm B | Group 4 Arm A | Group 4 Arm B
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/0 | 0/0 | 0/0 | 0/16 | 0/0 | 0/32 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/0 | 0/0 | 0/0 | 0/16 | 0/0 | 0/32 | 0/0
Other Adverse Events (participants affected / at risk) | 0/65 | 0/0 | 0/0 | 0/0 | 0/16 | 0/0 | 0/32 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated early and not powered for meaningful results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03187080/Prot_SAP_000.pdf